CLINICAL TRIAL: NCT00568555
Title: Effects of Low Dose Naltrexone in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: American Fibromyalgia Syndrome Association (Other)
Responsible Party: Principal Investigator, Sean Mackey, Associate Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SU-10232007-756; 8948
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Results first posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-09

CONDITIONS: Fibromyalgia; Persian Gulf Syndrome
MeSH Terms: conditions — Fibromyalgia; Persian Gulf Syndrome | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Low Dose Naltrexone first (Experimental): LDN first, then placebo.
  Interventions: Drug: Low Dose Naltrexone; Drug: Placebo - sugar pill
- Placebo - sugar pill first (Placebo Comparator): Placebo first, then LDN.
  Interventions: Drug: Low Dose Naltrexone; Drug: Placebo - sugar pill

INTERVENTIONS:
Drug: Low Dose Naltrexone — 3-4.5mg Naltrexone once daily
Drug: Placebo - sugar pill — Placebo pill once daily

SUMMARY:
Low Dose Naltrexone (LDN) has been reported anecdotally to reduce the symptoms of Fibromyalgia, a Chronic Multisystem Illness. The drug may work by regulating natural pain-reducing systems. In this study, we will administer both LDN and placebo to a small group of individuals with Fibromyalgia and Gulf War Syndrome, both Chronic Multisymptom Illnesses, to assess the drug's efficacy in treating the condition.

DETAILED DESCRIPTION:
This study will be a placebo-controlled, double-blind, cross-over drug tria. Patients with Primary Fibromyalgia or Gulf War Syndrome will be recruited from the Stanford University Pain Management Center and the surrounding community. Participation in the study will cover 22 weeks. Participants will attend a laboratory session 12 times for progress checkups, and will complete daily measures of symptoms.

ELIGIBILITY:
Inclusion Criteria:

Currently suffering from moderate to severe Fibromyalgia or symptoms of Gulf War Syndrome Age 18-65. Not taking any opioid analgesic Not pregnant or planning to become pregnant.

Exclusion Criteria:

Any known allergy to naltrexone or naloxone. Actual or planned pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jarred Younger, Sub-Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Younger J, Noor N, McCue R, Mackey S. Low-dose naltrexone for the treatment of fibromyalgia: findings of a small, randomized, double-blind, placebo-controlled, counterbalanced, crossover trial assessing daily pain levels. Arthritis Rheum. 2013 Feb;65(2):529-38. doi: 10.1002/art.37734. PMID 23359310

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 325 women completed an online web survey
Pre-assignment Details: Individuals were assessed for eligibility via web screening and phone screening prior to enrollment.
  Further eligibility (blood tests, questionnaires) assessed after enrollment; ineligible consented participants were withdrawn prior to assignment to groups.
Groups:
- Low Dose Naltrexone First: Low Dose Naltrexone (LDN) followed by placebo. LDN at 3-4.5mg, once a day. Placebo (sugar pill) once a day.
- Placebo - Sugar Pill First: Placebo first, followed by LDN. Placebo (sugar pill) once a day. LDN at 3-4.5mg, once a day.
Period: Overall Study
Arm/Group | Low Dose Naltrexone First | Placebo - Sugar Pill First
Started | 16 | 15
Completed | 15 | 14
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: 2 participants in the low dose naltrexone group did not have data to analyze (1 withdrew by patient choice, 1 had a malfunction with the data collection device)
  1 participant in the placebo condition did not have data to analyze (withdrew by patient choice)
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Naltrexone | Placebo - Sugar Pill | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (13.4) | 42.3 (13.0) | 42.7 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Pain Scores Between Baseline to End of Placebo Treatment and Between Baseline to End of LDN Treatment.
Description: Visual Analogue Scale for pain, 0 to 100, where 0=no pain and 100=worst pain imaginable.
  Baseline pain calculated averaging daily pain scores over the 2 week baseline period.
  Placebo and LDN pain scores calculated by averaging daily pain scores during the final 3 days of each condition.
  Values were converted to percent change in pain: [(baseline pain - end point pain)/baseline pain] x 100.
Time Frame: Baseline to end of placebo (2 weeks + 4 weeks) and baseline to end of LDN (2 weeks + 12 weeks)
Population: All completers
Measure: Mean (95% Confidence Interval); unit: percentage change from baseline to final
Groups:
- Low Dose Naltrexone: All participants during the Low Dose Naltrexone condition
- Placebo - Sugar Pill: All participants during the placebo condition
Arm/Group | Low Dose Naltrexone | Placebo - Sugar Pill
Number analyzed (Participants) | 28 | 28
percentage change from baseline to final | 28.8 [19.5 to 38.1] | 18.0 [7.2 to 28.8]

2. Secondary Outcome: Percent Change in Sleep Quality Scores Between Baseline to End of Placebo Treatment and Between Baseline to End of LDN Treatment.
Description: Visual Analogue Scale for sleep quality, 0 to 100, where 0 = "did not sleep well at all" and 100 = "slept extremely well".
  Baseline sleep quality calculated by averaging daily scores over the 2 week baseline period.
  Placebo and LDN sleep quality scores calculated by averaging daily scores during the final 3 days of each condition.
  Values were converted to percent change in sleep quality: [(baseline sleep - end point sleep)/baseline sleep] x 100.
Time Frame: Baseline to end of placebo (2 weeks + 4 weeks) and baseline to end of LDN (2 weeks + 12 weeks)
Population: All completers
Measure: Mean (95% Confidence Interval); unit: percentage change from baseline
Groups:
- Placebo - Sugar Pill: All participant during the placebo condition
Arm/Group | Low Dose Naltrexone | Placebo - Sugar Pill
Number analyzed (Participants) | 28 | 28
percentage change from baseline | 10.4 [-35.8 to 56.6] | 9.2 [-40.6 to 59]

3. Secondary Outcome: Percent Change in Fatigue Scores Between Baseline to End of Placebo Treatment and Between Baseline to End of LDN Treatment.
Description: Visual Analogue Scale for fatigue, 0 to 100, where 0 = "no fatigue at all" and 100 = "severe fatigue".
  Baseline fatigue calculated averaging daily scores over the 2 week baseline period.
  Placebo and LDN fatigue scores calculated by averaging daily scores during the final 3 days of each condition.
  Values were converted to percent change in fatigue: [(baseline fatigue - end point fatigue)/baseline fatigue] x 100.
Time Frame: Baseline to end of placebo (2 weeks + 4 weeks) and baseline to end of LDN (2 weeks + 12 weeks)
Population: All completers
Measure: Mean (95% Confidence Interval); unit: percentage change from baseline
Arm/Group | Low Dose Naltrexone | Placebo - Sugar Pill
Number analyzed (Participants) | 28 | 28
percentage change from baseline | 12.6 [-33.2 to 58.4] | 7.8 [-26.6 to 42.2]

4. Secondary Outcome: Percent Change in Pressure Pain Threshold Between Baseline and End of Placebo Treatment and Between Baseline to End of LDN Treatment.
Description: An algometer is used to apply pressure to 18 points across the body. Pressure is applied until the first sensation of pain in indicated. This pressure is recorded (as kg/cm2) and averaged for all 18 points to provide an overall score.
Time Frame: Baseline to end of placebo (2 weeks + 4 weeks) and baseline to end of LDN (2 weeks + 12 weeks)
Population: All completers
Measure: Mean (95% Confidence Interval); unit: percentage change from baseline to final
Arm/Group | Low Dose Naltrexone | Placebo - Sugar Pill
Number analyzed (Participants) | 28 | 28
percentage change from baseline to final | 36.70 [17.41 to 56.00] | 28.26 [11.27 to 45.24]

5. Secondary Outcome: Percent Change in Heat Pain Sensitivity Between Baseline and End of Placebo Treatment and Between Baseline to End of LDN Treatment.
Description: A thermode is placed on the palm, and temperature is increased until the first sensation of pain. That temperature is recorded in Degrees Celsius . The procedure is repeated 3 times and results are averaged into a single temperature recording.
Time Frame: Baseline to end of placebo (2 weeks + 4 weeks) and baseline to end of LDN (2 weeks + 12 weeks)
Population: All completers
Measure: Mean (95% Confidence Interval); unit: percentage change from baseline to final
Arm/Group | Low Dose Naltrexone | Placebo - Sugar Pill
Number analyzed (Participants) | 28 | 28
percentage change from baseline to final | 3.12 [0.40 to 5.83] | 3.45 [0.93 to 5.98]

ADVERSE EVENTS:
Arm/Group | Low Dose Naltrexone | Placebo - Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 20/28 | 7/28
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose Naltrexone (N=28) | Placebo - Sugar Pill (N=28)
Vivid Dreams (General disorders) | 10 | 4
Headache (General disorders) | 4 | 1
Nausea/Upset Stomach (General disorders) | 4 | 2
Nightmares (General disorders) | 3 | 1
Insomnia (General disorders) | 4 | 3
Dry mouth or throat (General disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No